CLINICAL TRIAL: NCT01590186
Title: Examination and Treatment of Pain in Front Foot
Status: Completed | Type: Observational
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Collaborators: Aalborg University Hospital (Other); Aalborg University (Other)
Responsible Party: Sponsor
Other Study IDs: ON-02-003-OSi
Record Dates: First submitted 2011-01-05; First posted 2012-05-02 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Pain
Keywords: Pain; Front foot; Flat foot; Metatarsalgia
MeSH Terms: conditions — Pain; Flatfoot; Metatarsalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
Tibial flat foot deformity is the most common reason for metatarsalgia. Flat foot deformity is a sign of degenerated problems such as weakness in ligament or fractures. Furthermore, metatarsalgia can be a sign of excessive load caused by sport activities or at work. The condition is very common at diabetics and patients with rheumatism.

The purpose of the study is to examine the load under the front foot at health people and patients with metatarsalgia. Furthermore, the researchers aim at being able to assess the best treatment of the flat foot deformity at each patient.

ELIGIBILITY:
Inclusion Criteria:

* Examination and treatment of pain in front foot

Exclusion Criteria:

* Normal gait
* No pains

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Examination and treatment of pain in front foot
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2002-10; Primary Completion 2003-04 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mogens B Laursen, MD, Principal Investigator — Northern Orthopaedic Division
Locations (1):
- Northern Orthopaedic Division, Clinic Aalborg, Aalborg, Northern Jutland, Denmark